CLINICAL TRIAL: NCT07098351
Title: A Clinical Study on the Efficacy and Safety of Nalfurafine Hydrochloride Orally Disintegrating Tablets in the Treatment of Moderate to Severe Pruritus in Peritoneal Dialysis Patients
Brief Title: Efficacy and Safety of Nalfurafine Hydrochloride ODT for Moderate-to-Severe Pruritus in Patients on Peritoneal Dialysis
Acronym: KARE-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSS-Remitch-PD-IIT-05
Record Dates: First submitted 2025-05-23; First posted 2025-08-01 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Adverse Event; Peritoneal Dialysis; Moderate-to-severe Pruritus; Chronic Kidney Disease-associated Itch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Singe-arm study: active treatment group (Other): Nalfurafine Hydrochloride Orally Disintegrating Tablets should be initially administered at a dose of 2.5 μg once daily after dinner or before bedtime for two consecutive weeks. After this initial treatment period, the dose should be adjusted based on the therapeutic response assessed by the change in Visual Analog Scale (VAS) scores for pruritus. If the treatment is effective, defined as a reduction of ≥20 mm in the average VAS score at Week 2 compared to baseline, the patient should continue taking 2.5 μg once daily for another two weeks. If the treatment response is inadequate (failure to meet the ≥20 mm VAS reduction criterion), the dose should be increased to 5 μg once daily and maintained for an additional two weeks. The medication should be taken consistently either after dinner or prior to bedtime throughout the treatment course.
  Interventions: Drug: Remitch

INTERVENTIONS:
Drug: Remitch — Nalfurafine 2.5μg daily for 2 weeks. Afterwards, the dose can be increased to 5μg daily if necessary (maximum dose not exceeding 5μg daily), continued for another 2 weeks.

SUMMARY:
Moderate to severe pruritus significantly impairs the quality of life in peritoneal dialysis patients, and effective treatment options remain limited. κ-opioid receptor agonists may alleviate itching by modulating neural signaling pathways. This study is a multicenter, prospective, single-arm clinical trial, planning to enroll 93 patients. It aims to test the hypothesis that nalfurafine hydrochloride orally disintegrating tablets compared to baseline, with acceptable safety.

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm clinical study designed to evaluate the efficacy and safety of nalfurafine hydrochloride orally disintegrating tablets in treating moderate-to-severe pruritus in peritoneal dialysis patients. The study consists of three phases: a screening period (1-2 weeks), a treatment period (4 weeks), and a follow-up period (1 week). During the screening phase, baseline pruritus levels are established using the Visual Analog Scale (VAS) and the Shichuan-Kawashima Pruritus Severity Score. The treatment period begins with an initial dose of 2.5 μg/day, which may be adjusted to 5 μg/day after 2 weeks based on symptom response; the follow-up phase assesses pruritus improvement and safety. The study plans to enroll 93 patients (including a 20% dropout rate), with the primary endpoint being the change in VAS score from baseline to week 4 of treatment. Secondary endpoints include VAS score changes at different stages, quality-of-life improvements, and adverse event incidence.

Eligible patients are aged 18-85 years, undergoing regular peritoneal dialysis for ≥3 months, and meeting baseline VAS criteria for moderate-to-severe pruritus. The primary efficacy measure is the mean change in daily maximum VAS scores (baseline vs. week 4), while secondary measures include pruritus severity scores, sleep quality, dose adjustment rates, and laboratory safety data. Statistical analyses will follow intention-to-treat (ITT) and per-protocol (PP) principles. Based on preliminary data (mean 28.4 mm, standard deviation 21.82 mm), the sample size calculation ensures 95% power to validate efficacy hypotheses.

The intervention involves monotherapy with nalfurafine hydrochloride orally disintegrating tablets, starting at 2.5 μg/day, with a potential increase to 5 μg/day after 2 weeks. Standardized scales assess pruritus, quality of life, and sleep improvements, alongside monitoring of vital signs, electrocardiograms, and laboratory parameters for safety evaluation. Enrollment criteria require ≥5 days of recorded morning/evening VAS scores during the baseline period (average ≥50 mm) and ≥2 days with Shichuan-Kawashima pruritus scores ≥3 (moderate severity).

The study anticipates a significant reduction in VAS scores as the primary endpoint, with secondary endpoints including dose adjustments, safety events, and patient-reported outcomes. This single-arm self-controlled study validates drug efficacy while strictly controlling dropout rates and data integrity to ensure result reliability.

ELIGIBILITY:
Inclusion Criteria:

At the time of signing informed consent:

* Aged 18-85 years (inclusive), regardless of gender.
* Chronic renal failure patients on regular peritoneal dialysis for ≥3 months, with no anticipated major treatment changes or rapid disease progression during the trial.
* Able to understand and comply with study procedures, voluntarily participate, and provide written informed consent.

At formal enrollment:

* During the baseline period, ≥5 days with both morning and evening VAS scores recorded, and the average of the higher VAS values (morning/evening) ≥50 mm.
* During the baseline period, ≥5 days with Xie-Kawashima itching severity assessed both morning and evening, including ≥2 days where the maximum itching score (morning/evening) was ≥3 (moderate).

Exclusion Criteria:

* Poor dialysis compliance, deemed by the investigator to affect efficacy/safety assessments.
* Poor dialysis compliance, deemed by the investigator to affect efficacy/safety assessments.
* Peritoneal dialysis regimen adjusted within 2 weeks prior to screening.
* Currently on or planning hemodialysis within 2 months.
* Planned kidney transplant or elective surgery during the study.
* Peritonitis within 4 weeks prior to screening, unable to continue peritoneal dialysis.
* ALT, AST, GGT, or total bilirubin >2× upper limit of normal (ULN) during screening.
* Pruritus not caused by chronic kidney disease (e.g., allergic, physical, infectious skin diseases, cholestatic liver disease).
* Severe cardiovascular disease (NYHA Class III/IV, acute MI, unstable angina, large pericardial effusion, severe arrhythmia, or ECG abnormalities deemed unsafe for participation).
* Active malignancy within 12 months prior to screening, or recent radiotherapy/chemotherapy/targeted/immunotherapy.
* Uncontrolled or drug-treated fungal/bacterial/viral infections (e.g., active TB, HIV).
* Uncontrolled hypertension (SBP ≥180 mmHg or DBP ≥110 mmHg).
* Current systemic corticosteroids/immunosuppressants (topical excluded).
* Psychiatric or cognitive disorders.
* Initiated/adjusted restricted medications (antihistamines, systemic/local corticosteroids [excluding ear/eye], calcineurin inhibitors, gabapentin, pregabalin) within 7 days prior to screening, or anticipated changes during the study.
* Initiated/adjusted medications affecting pruritus assessment (antipsychotics, hypnotics, SSRIs, anxiolytics, TCAs) within 2 weeks prior to screening, or anticipated changes during the study.
* Opioid agonists/antagonists used within 2 weeks prior to screening.
* Phototherapy for pruritus within 1 month prior to screening.
* History of drug abuse, dependence, or alcoholism within 12 months prior to screening.
* Allergy to opioids or trial drug excipients.
* Participation in another clinical trial with investigational drugs/devices within 28 days prior to screening, or residual investigational drug within 5 half-lives.
* Pregnant, breastfeeding, positive pregnancy test, or unwilling to use contraception during the study.
* Other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) score for Itch from baseline to Week4 of treatment period | This study includes a screening period (1-2 weeks, baseline assessment), a 4-week treatment phase (starting with nalfurafine 2.5μg/day, potentially increased to 5μg), and a 1-week follow-up period (to evaluate changes in itching severity).
  Calculation:
  Change = (Average of daily maximum VAS scores during baseline period) - (Average of daily maximum VAS scores during the 4th week of treatment period). Only dates with both daytime and nighttime VAS recordings were included in the assessment.
  Daily maximum VAS score:
  Defined as the higher value between the VAS measured at waking and bedtime each day.
  VAS scores range from 0 to 10 points.0 = "No itch" ,10 = "Worst itch". Higher scores indicate worse itch severity.

SECONDARY OUTCOMES:
Change in Visual Analog Scale(VAS) for Itch scores at Weeks 1, 2, 4 of treatment and follow-up period | Baseline, Week 1, Week 2, Week 4, and Follow-up
  Change from baseline in daily maximum Visual Analog Scale for Itch (VAS) scores at each assessment time point (Weeks 1, 2, 4 of treatment and follow-up period).VAS scores range from 0 to 10 points.0 = "No itch" ,10 = "Worst itch". Higher scores indicate worse itch severity.
Change in Xie-Kawashima Itch Scale scores | Baseline, Week 1, Week 2, Week 4, and Follow-up
  Change from baseline in daily maximum Xie-Kawashima Itch Scale scores at each assessment time point (Weeks 1, 2, 4 of treatment and follow-up period).
  Xie-Kawashima Itch Scale scores range from 0 to 4 points.0 = "No itch" ,4 = "Worst itch". Higher scores indicate worse itch severity.
The degree of change in Visual Analog Scale (VAS) scores from Baseline to Week 2,4 of treatment period | Baseline to Week 2,4 of treatment period
  Change of itch intensity,assessed by the Visual Analog Scale for Itch from baseline to Week 2,4 of treatment period.
  Calculated as: average of baseline VAS score minus average of VAS score during Week 2,4 of treatment period.
  Response Criteria:
  Clinically Significant Improvement:Mean VAS score < 20 mm during treatment period OR reduction ≥40 mm from baseline Improvement:Reduction ≥20 mm but <40 mm from baseline (excluding Clinically Significant Improvement) No Clinically Meaningful Improvement:Neither Category 1 nor Category 2 criteria met.
Change in Health-Related Quality of Life Scores | Baseline to Week 4 of treatment period
  Kidney Disease Quality of Life-36 (KDQOL-36) Scale score Range: 36-185 points.Higher scores indicate better quality of life.
  Skindex-16 Dermatology Life Quality Index Scale score Range: 0-96 points.Higher scores indicate worse quality of life.
Change in Pittsburgh Sleep Quality Index (PSQI) total score | Baseline to Week 4 of treatment period
  Change from baseline to Week 4 of treatment in sleep quality measured by Pittsburgh Sleep Quality Index (PSQI).
  Total Score Range: 0 to 21 points.Higher scores indicate worse sleep quality.
Proportion of participants escalating dosage of nalfurafine hydrochloride | Day 1 to Week 4 of treatment period
  Proportion of participants escalating dosage from 2.5μg QD to 5μg QD during 4-week treatment period.
  Drug Formulation: Nalfurafine hydrochloride orally disintegrating tablets.
  Calculation:
  Numerator: Patients with dose escalation Denominator: Total treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No